CLINICAL TRIAL: NCT05042310
Title: A Phase 1, Randomized, Participant- and Investigator-Blind, Placebo-Controlled, Single- and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3541860 in Healthy Japanese and Non-Japanese Participants
Brief Title: A Study of LY3541860 in Healthy Japanese and Non-Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18115; J3K-MC-KIAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-09-08; First posted 2021-09-13 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LY3541860 (Part A) (Experimental): Single doses of LY3541860 administered intravenously (IV) or subcutaneously (SC).
  Interventions: Drug: LY3541860
- LY3541860 (Part B) (Experimental): Multiple doses of LY3541860 administered either IV or SC.
  Interventions: Drug: LY3541860
- Placebo (Part A) (Placebo Comparator): Single doses of Placebo administered either IV or SC.
  Interventions: Drug: Placebo
- Placebo (Part B) (Placebo Comparator): Multiple doses of Placebo administered either IV or SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3541860 — Administered either IV or SC.
  Arms: LY3541860 (Part A); LY3541860 (Part B)
Drug: Placebo — Administered either IV or SC.
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3541860 in healthy Japanese and non-Japanese participants. The study will also assess how fast LY3541860 gets into the blood stream and how long it takes the body to remove it. The study is open to healthy participants. The study will last up to approximately 113 days.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female not of childbearing potential
* Have a body weight between 18 and 32 kilograms per square meter (kg/m²) and a body weight ≥ 50 kilograms (kg)
* Have veins suitable for blood sampling

Exclusion Criteria:

* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Have active or latent TB
* Have had breast cancer within the past 10 years or had lymphoma, leukemia, or any malignancy within the past 5 years
* Show clinical evidence of syphilis, HIV, hepatitis C, or hepatitis B, and/or test positive
* Have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing.
* Have previously completed a clinical trial investigating any other molecule targeting CD19, CD20 or have previously discontinued from this study after receiving LY3541860
* Are currently participating in or completed a clinical trial within the last 30 days
* Have received a vaccine containing a live (attenuated) virus within 28 days of screening or intend to receive during the course of the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 113
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3541860 | Predose on Day 1 through Day 113
  PK: Cmax of LY3541860
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3541860 | Predose on Day 1 through Day 113
  PK: AUC of LY3541860

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- P-One Clinic, Hachiōji, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No